CLINICAL TRIAL: NCT03942263
Title: KLIO - Non-interventional Multicenter Prospective and Retrospective Study to Describe Treatment Patterns and Disease Control in Patients With Classical Hodgkin's Lymphoma (cHL) and Systemic Anaplastic Large Cell Lymphoma (sALCL) in Routine Clinical Practice in the Russian Federation
Brief Title: A Study to Describe Treatment Patterns and Disease Control in Participants With cHL and sALCL in Routine Clinical Practice in the Russian Federation
Acronym: KLIO
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: CHL-5004; U1111-1229-0611 (Registry Identifier: WHO)
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Hodgkin Disease; Lymphoma, Large-cell, Anaplastic
Keywords: Drug Therapy
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newly Diagnosed and RR cHL Participants: Participants diagnosed with RR cHL at the time of enrollment and RR cHL within 3 years prior to inclusion in the study will be observed retrospectively. Participants with newly diagnosed cHL, or RR cHL at the time of enrolment, or RR cHL within 3 years prior to inclusion in the study will be observed prospectively for a period of 2 years. Data will be collected from 50 investigational sites to collect information on various treatment options, real-world effectiveness, outcomes and safety within the routine clinical setting.
- Newly Diagnosed and RR sALCL Participants: Participants diagnosed with RR sALCL at the time of enrollment and RR sALCL within 3 years prior to inclusion in the study will be observed retrospectively. Participants with newly diagnosed sALCL, or RR sALCL at the time of enrolment, or RR sALCL within 3 years prior to inclusion in the study will be observed prospectively for a period of 2 years. Data will be collected from 50 investigational sites to collect information on various treatment options, real-world effectiveness, outcomes and safety within the routine clinical setting.

SUMMARY:
The purpose of this study is to describe patterns of treatment used for cHL and sALCL in real world setting.

DETAILED DESCRIPTION:
This is a non-interventional, prospective and retrospective study of participants with cHL and sALCL. The study will collect information on therapy and outcome of cHL and sALCL in real-life clinical practice.

The study will enroll approximately 2000 participants. Based on the diagnosis of the disease, participants will be assigned to one of the following groups:

* Newly Diagnosed and RR cHL Participants
* Newly Diagnosed and RR sALCL Participants

This multi-center trial will be conducted in Russia. The retrospective data will be collected for the participants with RR cHL or RR sALCL at the time of enrollment and for participants with RR cHL or RR sALCL within 3 years prior to inclusion in the study at Visit 1 (Baseline). The prospective data will be collected for a period of 2 years from Visit 1 (Baseline) to Visit 5 (Month 24, Final Visit), both for newly diagnosed participants with cHL or sALCL and participants with RR cHL or RR sALCL at the time of enrolment, and participants with RR cHL or RR sALCL within 3 years prior to inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants 18 years or older by the time of enrollment.
2. Histologically confirmed diagnosis of cHL or sALCL.
3. Newly diagnosed participants, or participants with RR cHL or RR sALCL at the time of enrollment, or participants with RR cHL or RR sALCL within 3 years prior to inclusion in the Study.

Exclusion Criteria:

1. Unconfirmed diagnosis of cHL or sALCL.
2. Current, previous (within the last 3 years) or planned (for the next 2 years) participation in interventional clinical trials.
3. Participation in the non-interventional study CHL-5001 "An international, multi-centre, non-interventional retrospective study to describe treatment pathways, outcomes, and resource use in participants with classical Hodgkin lymphoma (B-HOLISTIC)" (Sponsor is Takeda Pharmaceuticals International AG).
4. Participants for whom the minimum study dataset was not available from their hospital medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with newly diagnosed cHL or sALCL, or with RR cHL or RR sALCL at the time of enrollment, or with RR cHL or RR sALCL within 3 years prior to inclusion in the study will be observed both retrospectively and prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Description of Treatment Patterns Used for cHL or sALCL | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Percentage of Participants Receiving Various Chemotherapy Regimens | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Percentage of Participants who Received Chemotherapy Regimens as per National Guidelines | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Percentage of Participants who Received Radiotherapy Including Site (Extended/Involved) and Total Dosing | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Percentage of Participants who Received Autologous Stem Cell Transplantation (AutoSCT) | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Percentage of Participants who Were Eligible for AutoSCT did not Receive it (Including Reasons) | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Percentage of Participants who Received Allogeneic Stem Cell Transplantation (AlloSCT) | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Distribution of Pre-SCT Therapy Regimens | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Distribution of First Line Treatment Patterns According to Prognostic Group | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Distribution of Relapse/Refractory (RR) Treatment Patterns | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)

SECONDARY OUTCOMES:
Overall Survival (OS) | From the date of cHL or sALCL diagnosis confirmation until the date of death from any cause or till the latest date of participant observed (up to Month 24)
  OS is defined as the time passed from the date of cHL or sALCL diagnosis confirmation until the date of death from any cause or till the latest date of participant observed.
Disease Free Survival-1 (DSF1) | From date of complete remission after first line of therapy up to relapse or till the latest date of participant observed (up to Month 24)
  DFS1 is defined as the time from the date of complete remission after first line of therapy till relapse or till the latest date of participant observed.
Freedom From Treatment Failure-1 (FFTF1) | From date of initiation first therapy until any treatment failures such as disease progression, not achieving complete remission after therapy, relapse, discontinuation of therapy for complications, death from any cause or till observed (up to Month 24)
  FFTF1 is defined as the time passed from date of initiation first therapy until any treatment failures such as disease progression, do not achieving complete remission after therapy, relapse, discontinuation of therapy for complications, death from any cause or till the latest date of participant observed.
Event Free Survival-1 (EFS1) | From date of initiation first therapy until therapy discontinuation, not achieving complete remission after therapy, progression, relapse, death from any cause, late therapy complications including second malignancies or till observed (up to Month 24)
  EFS-1 is defined as the time passed from date of initiation first line therapy until any events such as discontinuation of therapy for any reasons, do not achieving complete remission after therapy, progression, relapse, death from any cause, late therapy complications including second malignancies or till the latest date of participant observed.
Percentage of Participants with Complete Remission (CR) Achieved by the end of Treatment Regimen | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  CR based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 is defined as complete disappearance of all target lesions and all nodes with long axis less than (<) 10 millimeter (mm).
Percentage of Participants With Partial Remission (PR) Achieved by the end of Treatment Regimen | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  PR based on RECIST 1.1 is defined as greater than or equal to (>=) 30 percent (%) decrease in the sum of longest diameters (SLD) of target lesions but not a CR. CR is defined as complete disappearance of all target lesions and all nodes with long axis <10 mm.
Percentage of Participants With Overall Response Achieved by the end of Treatment Regimen | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  Overall response based on RECIST 1.1 is defined as the percentage of participants who have a PR or CR to therapy; it does not include stable disease and is a direct measure of drug tumoricidal activity. PR is defined as >=30% decrease in the SLD of target lesions but not a CR. CR is defined as complete disappearance of all target lesions and all nodes with long axis <10 mm.
Percentage of Participants With Stable Disease (SD) Achieved by the end of Treatment Regimen | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  SD based on RECIST 1.1 is defined as changes in the SLD of targeted lesions ranging between reduction of <10% to an increase by <20% without the appearance of a new lesion, and irrespective of positron emission tomography (PET) results.
Percentage of Participants With Progression Disease (PD) While on the Treatment | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  PD based on RECIST 1.1 is defined as >20% increase in the SLD of target lesions. For small lymph nodes measuring <15 mm post therapy, a minimum absolute increase of 5 mm and the long diameter should exceed 15 mm.
Percentage of Participants With Relapse (Both Early [<12 Months After the end of First Line Treatment] and Late Relapses) | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Percentage of Participants With Primary Resistance | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Percentage of Resistant Participants to the Second and Later Treatment Lines | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Percentage of Participants in Whom Brentuximab Vedotin was Used | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Distribution of Treatment Patterns Containing Brentuximab Vedotin in Clinical Practice | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Disease Free Survival (DFS) After the Treatment Line Including Brentuximab Vedotin Based on the Number of Cycles of Brentuximab Vedotin Performed Within this Treatment Line | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  DFS will be assessed after the treatment line including brentuximab vedotin based on the number of cycles of brentuximab vedotin performed within this Treatment Line. DFS is defined as the time from the date of complete remission till relapse or till the latest date of participant observed.
FFTF Based on the Number of Cycles of Brentuximab Vedotin Performed Within the Treatment Line | From initiation therapy date until any treatment failures such as disease progression, not achieving complete remission after therapy, relapse, discontinuation of therapy for complication, death from any cause, or till observed (up to Month 24)
  FFTF will be assessed based on the number of cycles of brentuximab vedotin performed within this treatment line. FFTF is defined as the time passed from date of initiation therapy until any treatment failures such as disease progression, do not achieving complete remission after therapy, relapse, discontinuation of therapy for complications, death from any cause or till the latest date of participant observed.
EFS Based on the Number of Cycles of Brentuximab Vedotin Performed Within this Treatment Line | From initiation therapy date until therapy discontinuation, not achieving complete remission after therapy, progression, relapse, death from any cause, late therapy complications including second malignancies or till observed (up to Month 24)
  EFS will be assessed based on the number cycles of brentuximab vedotin performed within this treatment line. EFS is defined as the time passed from date of initiation therapy until any events such as discontinuation of therapy for any reasons, do not achieving complete remission after therapy, progression, relapse, death from any cause, late therapy complications including second malignancies or till the latest date of participant observed.
Percentage of Participants With CR Achieved to the end of the Given Treatment Regimen Based on the Number of the Cycles of Brentuximab Vedotin Performed Within This Treatment Line | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  CR based on RECIST 1.1 is defined as complete disappearance of all target lesions and all nodes with long axis <10 mm.
Percentage of Participants With Overall Response Achieved to the end of the Given Treatment Regimen Based on the Number of the Cycles of Brentuximab Vedotin Performed Within This Treatment Line | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  Overall response is defined as the percentage of participants who have a partial or complete response to therapy; it does not include stable disease and is a direct measure of drug tumoricidal activity. PR is defined as >=30 % decrease in the SLD of target lesions but not a CR. CR is defined as complete disappearance of all target lesions and all nodes with long axis <10 mm.
Percentage of Participants With Progressive Disease Developed While on the Treatment Regimen Including Brentuximab Vedotin Achieved Based on the Number of the Cycles of Brentuximab Vedotin Performed Within This Treatment Line | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  PD based on RECIST 1.1 is defined as >20% increase in the SLD of target lesions. For small lymph nodes measuring <15 mm post therapy, a minimum absolute increase of 5 mm and the long diameter should exceed 15 mm.
Number of Cycles of Brentuximab Vedotin Before and After Stem Cell Transplantation (SCT) | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Distribution of Clinical Variables for cHL and sALCL at the Time of Primary Diagnosis | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  Clinical variable will include stage, histological types, immunohistochemistry data (yes/no), ALK-status (negative/positive), prognostic groups, prognostic risk factors (International Prognostic Score (IPS), International Prognostic Index, Age-adjusted International Prognostic Index, International T-cell Lymphoma Project Score, Prognostic Index for peripheral T-cell lymphoma unspecified [PTCL-U] [PIT]), prognostic risk factors, and risk factors for relapse.
Distribution of Clinical Variables for cHL and sALCL at the Time of Resistance/Relapses | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  Clinical variable will include stage, histological types, immunohistochemistry data (yes/no) and ALK-status (negative/positive).
Percentage of Participants for Whom PET and PET/Computed Tomography (CT) was Used for Primary Disease Diagnostic and Staging | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Percentage of Participants for Whom PET and PET/CT Scan was Used for Interim Treatment Response Evaluation | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
OS Based on use of PET/CT Scan for Initial Disease Staging, Interim and Final Response Assessment During Frontline and Second Line Treatment | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  OS is defined as the time passed from the date of initiation of cHL or sALCL treatment until the date of death from any cause or till the latest date of participant observed. OS will be analyzed by Cox regression.
Timepoint of Performing Interim Response Evaluation With PET/CT Scan (Number of Cycle After Which the Evaluation is Performed, Time From the Start of Last Cycle of Therapy) | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  Timepoints will include number of cycle after which the evaluation is performed and time from the start of last cycle of therapy.
Percentage of Participants for Whom PET and PET/CT Scan Were Used to Evaluate Final Treatment Response | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Timepoint of Performing Final Response Evaluation With PET/CT scan (Number of Cycle After Which the Evaluation is Performed, Time From the Start of Last Cycle of Therapy) | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  Timepoints will include number of cycle after which the evaluation is performed and time from the start of last cycle of therapy.
Time of Performing PET and PET/CT Scan After SCT | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Distribution of Imaging Patterns Used for Primary Disease Diagnostic and Staging in Different Regions of Russia | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Distribution of Imaging Patterns Used for Treatment Response Evaluation | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Distribution of Imaging Patterns Used for Disease Control of the Participants Being in Remission | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Percentage of cHL or sALCL Participants who Used Healthcare Resources: Hospitalizations, Sick Leave Sheet | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
  Healthcare resources will include hospitalizations and sick leave sheet.
Number of Hospitalizations | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Number of Days Spent on Hospital Beds | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Number of Sick Leaves | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Number of Days Spent on Sick Leaves | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)
Disease Free Survival-2 (DSF2) | From date of complete remission after second line of therapy up to relapse or till the latest date of participant observed (up to Month 24)
  DFS2 is defined as the time from the date of complete remission after second line of therapy till relapse or till the latest date of participant observed.
Freedom From Treatment Failure-2 (FFTF2) | From date of initiation second therapy until any treatment failures such as disease progression, not achieving complete remission after therapy, relapse, discontinuation of therapy for complications, death from any cause or till observed (up to Month 24)
  FFTF2 is defined as the time passed from date of initiation second line therapy until any treatment failures such as disease progression, do not achieving complete remission after therapy, relapse, discontinuation of therapy for complications, death from any cause or till the latest date of participant observed.
Event Free Survival-2 (EFS2) | From date of initiation second therapy until therapy discontinuation, not achieving complete remission after therapy, progression, relapse, death from any cause, late therapy complications including second malignancies or till observed (up to Month 24)
  EFS-2 is defined as the time passed from date of initiation second line therapy until any events such as discontinuation of therapy for any reasons, do not achieving complete remission after therapy, progression, relapse, death from any cause, late therapy complications including second malignancies or till the latest date of participant observed.
Number of Cycles of Brentuximub Vedotin Administered in Routine Clinical Practice | From frontline treatment for newly diagnosed participants or within 3 years prior to inclusion in the study for RR cHL or RR sALCL participants till end of participant observation in scope of the study (approximately 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (50):
- Russia (50):
  - State budgetary healthcare institution of the Astrakhan region Alexander-Mariinsky regional clinical hospital, Astrakhan
  - Autonomous Institution "Republican Clinical Oncology Dispensary" of the Ministry of Health of Chuvashia, Cheboksary
  - State budgetary health care institution "Chelyabinsk Regional Clinical Center for Oncology and Nuclear Medicine", Chelyabinsk
  - State Budget Public Health Institution "Regional Oncological Dispensary", Irkutsk
  - Kaluga Regional Clinical Oncologic Dispensary, Kaluga
  - Tatarstan Regional Clinical Cancer Center, Kazan'
  - State budgetary institution of health care of the Kemerovo region "Regional Clinical Oncology Center", Kemerovo
  - Regional State Budgetary Institution of Health "Regional Clinical Hospital 1" named after Professor S.I. Sergeeva, Ministry of Health of the Khabarovsk Territory, Khabarovsk
  - Federal State Budgetary Institution of Science "Kirov Research Institute of Hematology and Blood Transfusion of the Federal Medical and Biological Agency", Kirov
  - Regional State Budgetary Institution of Health "Kostroma Oncological Dispensary", Kostroma
  - Regional State Budgetary Institution of Health "Regional Clinical Hospital", Krasnoyarsk
  - Regional State Budgetary Institution of Healthcare Krasnoyarsk Regional Clinical Oncologic Dispensary named after A.I. Kryzhanovsky", Krasnoyarsk
  - Public health institution Lipetsk Regional Oncology Center, Lipetsk
  - State budgetary health care institution "Regional Oncology Center 2", Magnitogorsk
  - Federal State Budgetary Institution "Main Military Clinical Hospital named after Academician N.N.Burdenko" of the Ministry of Defense of the Russian Federation, Moscow
  - Federal State Budgetary Institution "National Medical-Surgical Center named after N.I. Pirogov" Ministry of Health of the Russian Federation, Moscow
  - Federal State Budgetary Institution "National Medical Research Center of Oncology named after N.N. Blokhina "of the Ministry of Health of the Russian Federation, Moscow
  - The Moscow State Clinical Hospital No. 52 of the Moscow City Department of Healthcare, State Budgetary Institution of Health Care, Moscow
  - Federal State Institution National Medical Research Center of Hematology of the Ministry of Health of the Russian Federation, Moscow
  - Moscow City Hematology Center on the basis of the State Budgetary Institution of Healthcare of the City of Moscow City Clinical Hospital named after S.P. Botkin Moscow Department of Health, Moscow
  - State Budgetary Institution of Healthcare of the Moscow Region Moscow Regional Research Clinical Institute named after M.F. Vladimirskoye, Moscow
  - State Budgetary Healthcare Facility of Nizhny Novgorod Region "City Clinical Hospital 12", Nizhny Novgorod
  - State budgetary institution of health care of the Nizhny Novgorod region "Regional Clinical Hospital named after NA Semashko", Nizhny Novgorod
  - State Budgetary Institution of Healthcare of the Novosibirsk Region "City Clinical Hospital No. 2", Novosibirsk
  - Federal State Budgetary Institution of Public Health of the Novosibirsk Region "Research Institute of Fundamental and Clinical Immunology", Novosibirsk
  - State Budgetary Institution of Healthcare of the Novosibirsk Region "State Novosibirsk Regional Clinical Hospital", Novosibirsk
  - Medical Radiological Research Center. A.F. Tsyba - a branch of the Federal State Budgetary Institution "Scientific Medical Research Center of Radiology" of the Ministry of Health of the Russian Federation, Obninsk
  - Budget institution of healthcare of Omsk region "Clinical Oncologic dispensary", Omsk
  - State budgetary institution of public health "Orenburg regional clinical hospital 1", Orenburg
  - The State Budgetary Institution of Healthcare "Regional Oncologic Dispensary", Penza
  - State Budgetary Institution of Healthcare of the Republic of Karelia Republican Hospital named after V. A. Baranova ", Petrozavodsk
  - State Budgetary Institution of Healthcare "Pskov Regional Clinical Oncologic Dispensary", Pskov
  - Federal State Budgetary Educational Institution of Higher Education Rostov State Medical University of the Ministry of Health of the Russian Federation, Rostov-on-Don
  - Federal State Budgetary Educational Institution of Higher Education Ryazan State Medical University named after Academician I.P. Pavlova" of the Ministry of Health of the Russian Federation, Ryazan
  - Federal State Budgetary Educational Institution of Higher Education "North-Western State Medical University named after II Mechnikov" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Federal State Budgetary Institution "Russian Research Institute of Hematology and Transfusiology of the Federal Medical and Biological Agency", Saint Petersburg
  - Federal State Budgetary Institution "N. N. Petrov National Medical Research Center of Oncology" of the Ministry of Health of Russia, Saint Petersburg
  - State Budgetary Institution of Healthcare Leningrad Regional Clinical Hospital, Saint Petersburg
  - Saratov State Medical University named after V.I.Razumovsky of the Ministry of Health of Russia "Clinic of Physiopathology and Hematology named after Professor V.Ya. Shustov", Saratov
  - Study State Budgetary Institution of Health "Oncology Dispensary No. 2" of the Ministry of Health of the Krasnodar Territory, Sochi
  - State Budgetary Institution of Healthcare of the Stavropol Territory "Stavropol Regional Clinical Oncology Dispensary", Stavropol
  - Budgetary institution of the Khanty-Mansiysk Autonomous Okrug Ugra, Surgut
  - State institution of the Komi Republic "Komi Republican Oncological Dispensary", Syktyvkar
  - State Healthcare Institution of Tula Region "Tula Regional Clinical Hospital", Tula
  - State autonomous health care institution of the Tyumen region "Multidisciplinary clinical medical center "Medical City", Tyumen
  - Ministry of Health of the Republic of Bashkortostan State Autonomous Healthcare Institution Republican Clinical Oncologic Dispensary, Ufa
  - State Healthcare Institution "Regional Clinical Oncologic Dispensary", Ulyanovsk
  - State budgetary health care institution "Volgograd Regional Clinical Oncology Center", Volgograd
  - Budget institution of health care of the Vologda region "Vologda regional clinical hospital", Vologda
  - State budgetary institution of health care of the Yaroslavl region "Regional Clinical Hospital", Yaroslavl

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603b4db2bf003ab4a2e1??page=1&idFilter=CHL-5004